CLINICAL TRIAL: NCT01563575
Title: WHO-HPH Recognition Project on Fast-Track Implementation of Clinical Health Promotion - a Multi-Centre RCT
Brief Title: WHO-HPH Recognition Project on Fast-Track Implementation of Clinical Health Promotion
Acronym: RP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: World Health Organization (Other); International Network of Health Promoting Hospitals & Health Services (HPH) (Unknown); National HPH Network of Montreal, Canada (Unknown); National HPH Network of the Czech Republic (Unknown); National HPH Network of Slovenia (Unknown); National HPH Network of Estonia (Unknown); Regional HPH Network of Taiwan (Unknown); National HPH Network of Indonesia (Unknown); National HPH Network of Japan (Unknown); HPH member hospitals in Denmark (Unknown); HPH member hospitals in Croatia (Unknown); HPH member hospitals in Malaysia (Unknown); HPH member hospitals in Thailand (Unknown)
Responsible Party: Principal Investigator, Hanne Tonnesen, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WHOHPHRP
Record Dates: First submitted 2012-03-22; First posted 2012-03-27 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Smoking; Excessive Drinking; Lack of Physical Activity; Malnutrition; Obesity
Keywords: Recognition Process; Health Promotion; HPH; WHO; Hospitals; Health Services; Health Gain; Service Delivery; Quality Management
MeSH Terms: conditions — Smoking; Sedentary Behavior; Malnutrition; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): fast-track implementation process
  Interventions: Other: fast-track implementation process
- Control Group (No Intervention): Continue usual routine

INTERVENTIONS:
Other: fast-track implementation process — Undergo fast-track implementation process (WHO-HPH recognition Process), including: baseline data collection, quality plan, implementation for one year, follow-up data collection, revision of quality plan, external site visit and data validation
  Arms: Intervention Group

SUMMARY:
The project's background is the notion that patient centred clinical health promotion has been shown to significantly improve both outcomes and patient safety. Accordingly, the WHO describes health promotion as a key dimension of quality in hospitals, and the organization has developed standards on the topic in order to help hospital management and staff members to assess and improve the quality of health care and thereby achieve better health for patients, staff, and community. Even so, however, health promotion is still a very implicit part of nearly all quality standards on hospitals. Moreover, assessing hospitals departments' health promotion performance is still quite an unexplored area. On this basis, this project will test a new recognition process that uses the relevant WHO-HPH tools and standards to assess performance, by way of explicit documentation and evaluation of clinical health promotion activity. The project is deigned as a RCT, with a control group that undergoes the recognition process immediately and a control group that continue usual clinical routine. Then, after one year, the control group also begins the recognition process (= delayed start), while the Intervention group (=immediate-start) continues with the recognition process. Doing this allows for a great array of measurements, and hopefully the project will then show whether the recognition process really benefits implementation of health promotion in hospitals and health services, and also, if this really generates better health gains for patients and staff. The outcome measurements will be frequency of health promotion services delivered on smoking, excessive alcohol use, overweight, malnutrition, and physical activity to patients in need. Such services could for instance be motivational counselling and brief interventions, as well as intervention, rehabilitation and after treatment. Physical, mental, and social health status among patients and staff will be measured by short form (SF36).

ELIGIBILITY:
Inclusion Criteria:

* Clinical hospital departments from university hospitals
* Clinical hospital departments from non-university hospitals

Exclusion Criteria:

* Palliative care departments
* Pediatric departments
* Nursing homes
* Non-hospital departments
* Primary care facilities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Changed health gain of patients and staff | Baseline, after 1 year, after 2 years
  Change in physical, mental, and social health status among patients and staff will be measured by short form (SF36).

SECONDARY OUTCOMES:
Number of health promotion services delivered | Baseline, after 1 year, after 2 years
  Change in the frequency of health promotion services delivered on smoking, excessive alcohol use, overweight, mal-nutrition, and physical activity to smoking, excessive drinking, overweight, malnourished, and physical inactive patients. These services concern clinical health promotion activities, like motivational counselling and brief interventions, as well as intervention, rehabilitation and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Tonnesen, MD DMSc, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (11):
- National HPH Network of Montreal, Canada, Montreal, Canada
- HPH Members in croatia, Zagreb, Croatia
- National HPH Network of the Czech Republic, Prague, Czechia
- HPH Members in Denmark, Middelfart, Denmark
- National HPH Network of the Estonia, Tallinn, Estonia
- National HPH Network of Indonesia, Jakarta, Indonesia
- National HPH Network of Japan, Tokyo, Japan
- HPH members in Malaysia, George Town, Pulau Pinang, Malaysia
- National HPH Network of Slovenia, Golnik, Slovenia
- Regional HPH Network of Taiwan, Taipei, Taiwan
- HPH members in Thailand, Bangkok, Thailand

REFERENCES:
- [Derived] Svane JK, Chiou ST, Groene O, Kalvachova M, Brkic MZ, Fukuba I, Harm T, Farkas J, Ang Y, Andersen MO, Tonnesen H. A WHO-HPH operational program versus usual routines for implementing clinical health promotion: an RCT in health promoting hospitals (HPH). Implement Sci. 2018 Dec 22;13(1):153. doi: 10.1186/s13012-018-0848-0. PMID 30577871
- See also: Main info page — http://www.hphnet.org/index.php?option=com_content&view=article&id=1954&Itemid=218